CLINICAL TRIAL: NCT04535635
Title: A Feasibility Study for a Randomized Control Trial of the Effects of Active Release Techniques® on Pain and Function of Lower Limb Myofascial Injuries
Brief Title: Effects of ART® on Lower Limb Myofascial Pain and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Memorial Chiropractic College (Other)
Responsible Party: Principal Investigator, Jason Pajaczkowski, Associate Professor, Canadian Memorial Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 192031
Record Dates: First submitted 2020-05-27; First posted 2020-09-02 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Muscle Injury; Lower Limb Injury
Keywords: myofascial pain syndromes; Active Release Techniques®; soft tissue therapy
MeSH Terms: conditions — Leg Injuries; Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: This study will consist of two groups - one receiving ART® and the other receiving a sham. Prior to the start of the study, an independent party (Dr. Lesley Bainbridge, Associate Professor at the University of British Columbia Department of Physical Therapy, Faculty of Medicine) will perform a two-group block randomization to determine which participants will receive the sham and which will receive ART®. The assessors, Mike Edgar and Frank Astri, will be blinded to the randomization and treatment allocation. The PI, Jason Pajaczkowski, will be blinded to the randomization process but as the treating clinician, he will know into which group each new participant has been allocated only at the time of presentation when he is required to open the next allocation sequence.
  The ART® procedure will consist of identifying and treating manipulatable lesions as per their protocols, while the sham group will receive a passable version of this technique.
Who Masked: Participant, Outcomes Assessor
Masking Description: An independent party (Dr. Lesley Bainbridge, Associate Professor at the University of British Columbia Department of Physical Therapy, Faculty of Medicine) will perform a two-group block randomization prior to the start of the trial. The PI will record clinical notes as per standards and include the group (ART or sham) in these notes. These notes are kept on a password-protected laptop that only he has access to. The assessors, Mike Edgar and Frank Astri, will be blinded to the randomization scheme and allocation. The participants will also be blinded to which group they are part of.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Techniques® (Experimental): The ART® procedure will consist of identifying and treating manipulatable lesions as per their protocols, while the sham group will receive a passable version of this technique. This information is under copyright and cannot be copied or outlined specifically in any form, including a research paper. The overarching procedure used by ART® will be explained however specific details referring to each protocol cannot be described. Muscles are shortened, and the therapist applies sufficient digital pressure to be in contact with the tissue in question. Directional tension is applied proximally along the muscle fiber direction, and then the structure is lengthened while the contact remains as described.
  Interventions: Other: Active Release Techniques®
- Sham Active Release Techniques® (Placebo Comparator): For the sham treatment, the muscle(s) in question will be taken from a lengthened to a shortened position (opposite of the protocol direction as per the ART® manual) with a broad light contact on the skin - the treating therapist will not achieve tissue depth as specified by ART® and will not attempt to take "tension" as is outlined in the ART® manual.
  Interventions: Other: Sham Active Release Techniques®

INTERVENTIONS:
Other: Active Release Techniques® — The ART® procedure will consist of identifying and treating manipulatable lesions as per their protocols, while the sham group will receive a passable version of this technique. This information is under copyright and cannot be copied or outlined specifically in any form, including a research paper. The overarching procedure used by ART® will be explained however specific details referring to each protocol cannot be described. Muscles are shortened, and the therapist applies sufficient digital pressure to be in contact with the tissue in question. Directional tension is applied proximally along the muscle fiber direction, and then the structure is lengthened while the contact remains as described.
  Arms: Active Release Techniques®
Other: Sham Active Release Techniques® — For the sham treatment, the muscle(s) in question will be taken from a lengthened to a shortened position (opposite of the protocol direction as per the ART® manual) with a broad light contact on the skin - the treating therapist will not achieve tissue depth as specified by ART® and will not attempt to take "tension" as is outlined in the ART® manual.
  Arms: Sham Active Release Techniques®

SUMMARY:
This is a feasibility study to determine if the investigators can conduct a clinical trial with a sham and control soft tissue treatment. The primary research questions are can the investigators provide the treatments as specified, can they recruit a sufficient number of participants, and does ART® decrease pain and improve function in 20-50 year-old adults with subacute or chronic lower limb soft-tissue injuries compared to a sham treatment? This is a pre-post ART® pilot study with a control group that would receive a sham ART® treatment. The study group is 20-50 year-old adults with subacute or chronic lower limb soft tissue injuries.

DETAILED DESCRIPTION:
Active Release Techniques® (ART®) is amongst the most widely utilized soft tissue techniques in the world. It is estimated that the 15,000 practitioners that have been certified in ART®, a list that includes medical doctors, chiropractors, physiotherapists, athletic therapists, and massage therapists, have collectively provided approximately 22 million treatments 41. In addition to a wealth of anecdotal information, there are numerous papers, albeit of differing scientific rigor, aimed at substantiating these claims. The principal investigator and co-investigator have authored a systematic review on all the available published research concerning ART® (currently seeking publication). The paucity of quality research in and of itself is the reason the authors have recently completed a systematic review on ART. The lack of quality studies begs the question for future research to determine its efficacy. Common issues in the existing research include: lack of sample size calculation 14,20,28,34,48,50,54,55,59, lack of control group 6,14,20,28,50,53,54,55,59, lack of certified ART® providers 6,21,22,28,34,37,48,50,59,66 lack of identifiable manipulatable lesions14,20,21,28,48,50,59, poor inclusion/exclusion criteria 34,48,50, inappropriate outcome measures14,20,48,59, the use of asymptomatic study participants14,21,23,59, descriptive instead of inferential statistics 55,59, and using ART® for purposes other than which it was intended 20,21,22,48,50,59. This study being proposed will address all of these factors.

Current evidence supports that the palpatory sensation of fascia softening or lengthening is not the result of actual elongation in the fascial sheet itself. This is because the requisite forces to lengthen these dense fasciae far exceed the capacity of what can be generated therapeutically according to Chaudry et al.7. As per Schleip, a more plausible mechanism is that via neurological feedback, muscles in series with the fascia being treated are relaxing, thereby producing the sensation of a myofascial release 56. These potential changes in tissue stiffness and elasticity have never been studied following a course of ART® treatments. Elastography has been used to measure changes in tissue stiffness following massage however, at present ART® has yet to be studied using this modality. The Principal Investigator is currently working on a joint proposal with Central Queensland University in Australia to produce the first study in this field.

Sports chiropractors and athletes alike describe the benefit of Active Release Techniques® however, the current state of the literature is inconclusive, neither supporting nor refuting its effects. No studies to date have explored the relationship between the neuromuscular effects of ART® on the lower extremity in subacute myofascial pain with performance outcomes in 20-50 year-old adults. This study will contribute to the current literature on ART® and myofascial pain and performance in athletes, as well as the effect of ART® in symptomatic populations. This research adds to the body of research on one of the most widely used modalities in sports medicine and manual therapy. This study will further the work by Schleip by measuring lower limb neuromuscular function after ART® treatments. In addition, by using measures relating to motor control and pain, neuromuscular control becomes a construct of performance, where these findings can subsequently be applied to athletes and sports, particularly those involving running, jumping, and kicking. However, the results have implications for vocational endeavours as well and those experiencing lower limb discomfort. Riel et al found that the prevalence and incidence rates were 16.6 and 7.9 per 1000 registered patients respectively in general practice, so lower limb myofascial injuries are prevalent in non-athletic populations as well 61.

This pilot study will be, along with the author's publication of a systematic review of ART®, the cornerstone for proof of concept in obtaining funding for a large-scale clinical trial. The intent is to continue studying the efficacy of ART® across various conditions and athletic populations, while simultaneously beginning research on the mechanism by which ART® and all manual therapies affect their response.

ELIGIBILITY:
Inclusion Criteria:

* Any adult 20-50 years with a subacute or chronic lower myofascial injury
* Palpatory findings of a tight and tender area with a manipulatable lesion that reproduces the chief complaint (may include active vs latent trigger point)

Exclusion Criteria:

* Neurological conditions
* Degenerative joint disease of the lower limb
* Previous surgery in the area

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Change in the Lower Extremity Functional Scale | This outcome measure will be used to measure the change in disability. It will be collected twice - once during the intake (prior to beginning ART® or sham) as a baseline, and then a second time following the fourth (final) treatment 2 weeks later.
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress, and outcome, as well as to set functional goals.
  The LEFS can be used to evaluate the functional impairment of a patient with a disorder of one or both lower extremities. It can be used to monitor the patient over time and to evaluate the effectiveness of an intervention. The LEFS is graded on an 80 point scale (score can be between 0 and 80), where a lower number equates with less disability and higher number with more disability.

SECONDARY OUTCOMES:
Change in the Numeric Pain Rating Scale | This outcome measure will be used to measure the change in pain intensity. It will be collected twice - once during the intake (prior to beginning ART® or sham) as a baseline, and then a second time following the fourth (final) treatment 2 weeks later.
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). It has been shown that a composite scoring system including best, worse, and current level of pain over the last 24 hours was sufficient to pick up changes in pain intensity with maximal reliability. This is a 10-point scale, and the values can be any whole number between 0 and 10. Lower scores equate to less pain intensity, while higher scores indicate more pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Pajaczkowski, DC, Principal Investigator — Associate Professor, Canadian Memorial Chiropractic College
Locations (2):
- Canada (2):
  - SWAT Health, Mississauga, Ontario
  - Canadian Memorial Chiropractic College Main Campus Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
We are considering sharing the data we collected, although it will all be contained within the study itself. We will consult our research chair at the Canadian Memorial Chiropractic College for advisement.